CLINICAL TRIAL: NCT00592189
Title: Fetal Membrane as a New Coverage Material
Brief Title: Study of Donated Amnion, Fetal Placental Membrane, as Skin Substitute for Burn Patients
Acronym: Amnion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1999-209; Clayton
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Wounds
Keywords: Burns; Wound healing; Amnion
MeSH Terms: conditions — Wounds and Injuries; Burns | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Amnion tissue and blood collection
  Interventions: Procedure: blood draw

INTERVENTIONS:
Procedure: blood draw — blood collection

SUMMARY:
Is the use of fetal membrane (human amnion) as a transient wound coverage in wound repair safe and efficacious.

Will the incorporation of liposomal gene constructs to amnion enhance the functionality of human amnion and improve wound repair.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Pregnant, delivery expected within the month

Exclusion Criteria:

* Known history of hepatitis, HIV, or active transmissable diseases

Ages: 16 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1164 (Actual)
Dates: Start 1999-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Safe method of obtaining and processing amnion | 0-21 days post harvest

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States